CLINICAL TRIAL: NCT05221593
Title: Evaluation of Lithium Efficacy Against Chemotherapy Induced Neutropenia in Breast Cancer Patients
Brief Title: Efficacy of Lithium Against Chemotherapy Induced Neutropenia in Breast Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed osama elbastawesy hassan elkasar, Principal Investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: lithium and breast cancer
Record Dates: First submitted 2021-12-25; First posted 2022-02-03 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Neutropenia
MeSH Terms: conditions — Neutropenia | interventions — Lithium Carbonate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (No Intervention): will receive chemotherapy regimen with placebo
- study group (Experimental): will receive chemotherapy regimen with Lithium Carbonate in controlled release formula (400mg b.i.d).
  In order to avoid the potential for bone marrow stimulation at the time chemotherapy was administered, the administration of lithium was started 24 hours after the administration of chemotherapy and continued for 18 days of every 21.the lithium serum level will be measured at specific times to ensure lithium serum level between 0.4-0.8 mmol\L along the treatment course.
  Interventions: Drug: Lithium Carbonate

INTERVENTIONS:
Drug: Lithium Carbonate — 400 mg tablet in controlled released formula
  Other Names: Prianil controlled-release tablet
  Arms: study group

SUMMARY:
Using Lithium Carbonate to decrease incidence of neutropenia caused by using chemotherapy regimen in breast cancer patients.

DETAILED DESCRIPTION:
Introduction:

Cytotoxic chemotherapy predictably suppresses the hematopoietic system, impairing host protective mechanisms. Neutropenia is the most serious hematologic toxicity of cancer chemotherapy, often limiting the doses of chemotherapy that can be tolerated. The degree and duration of the neutropenia determine the risk of infection. The Common Toxicity Criteria of the National Cancer Institute is the most commonly used scale for grading the severity of the cytopenias associated with cancer chemotherapy; it delineates neutropenia into 4 grades. Chemotherapy predisposes patients with cancer to infections both by suppressing the production of neutrophils and by cytotoxic effects on the cells that line the alimentary tract. Neutrophils are the first line of defence against infection as the first cellular component of the inflammatory response and a key component of innate immunity. Neutropenia blunts the inflammatory response to nascent infections, allowing bacterial multiplication and invasion. Because neutropenia reduces the signs and symptoms of infection, patients with neutropenia often may present with fever as the only sign of infection. In this setting, patients with fever and neutropenia, or febrile neutropenia (FN), must be treated aggressively, typically with intravenous antibiotics and hospitalization, because of the risk of death from rapidly spreading infection. The availability of hematopoietic growth factors and improvements in antibiotic therapy have changed greatly how clinicians approach the management of neutropenia, yet this complication remains a central concern in the delivery of cancer chemotherapy.

Lithium carbonate continues to be the most useful agent available for the prophylaxis and treatment of bipolar illness. Lithium augmentation of antidepressants is useful in the treatment of resistant unipolar depression. Its utility in other psychiatric disorders such as schizophrenia, alcoholism, or aggressive behaviour is documented only when a significant affective component exists. Hematologic changes have been associated with lithium Unexplained increases in white blood cell (WBC) counts have occurred in psychiatric patients treated with lithium. This leukocytosis occurs within 1 week of treatment and is reversible. It is unrelated to age, sex, or diagnosis. Although serum levels above 0.5 milliequivalent/L are required for the effect, there is no proportional response to dose. In 1998, Ballin et al prospectively examined eight adult patients with bipolar disorder to find whether lithium carbonate increased their peripheral blood cluster of differentiation 34 (CD34) hematopoietic stem cells (HSC). The administration of lithium salts to haematologically normal subjects is associated with increased marrow neutrophil production and enhanced release of granulocyte colony stimulating factor (G-CSF) in vitro, followed by peripheral blood neutrophilia.The unsaturated vitamin B12-binding capacity, an indirect assessment of the total-body granulocyte pool, is elevated in patients taking lithium for manic-depressive psychosis. In man, oral lithium carbonate raises urinary levels of G-CSF and augments production of G-CSF by peripheral blood mononucleated cell. Moreover, when Levitt and Quesenberry studied the effects of adding lithium to a murine bone marrow liquid culture system, lithium substantially increased the number of granulocyte-committed progenitor cells and pluripotential stem cells. Lithium therefore seems to have at least two distinct actions in haematopoiesis: It enhances the production of G-CSF, and it directly stimulates the proliferation of pluripotential stem cells. In 1978, Stein et al. first formally showed that lithium-induced granulocytosis was not merely a redistribution of granulocytes that are marginated or are in the marrow reserves, supporting the hypothesis of increased granulocyte production. Lithium also affects cytokines that involved in mobilization of neutrophils from bone marrow to blood through inhibition of Glycogen synthase kinase 3 (GSK-3) function, thereby indirectly increasing the attractive CXCL12 gradient toward a hypoxic marrow trophic niche, where HSCs can thrive. This is reflected by increased marrow trophic niche function: peripheral neutrophilia, increased platelets, and increased CD34+ counts.

Additionally, lithium has anticancer activity and neuroprotective properties. One piece of experimental evidence for lithium's potential as a cancer therapy is that inhibition of GSK3 was observed to inhibit prostate cancer cell proliferation. With respect to colorectal cancer, it has been found that lithium inhibits proliferation of a colorectal cancer cell line. Phosphatase and tensin homolog (PTEN) overexpression and lithium administration were shown to cooperatively inhibit proliferation of colorectal cancer cells. Because lithium therapy is systemic rather than topical or local, it follows that lithium might inhibit metastasis. Evidence that this is the case for colon cancer comes from observation of inhibition of metastasis-inducing factors by lithium and by observation on reduced metastasis in model animals given lithium therapy. Autophagy is a key cellular process in the inhibition of cancer. Lithium has been shown to induce autophagy, due to its inhibition of inositol monophosphatase.

For these issues that mentioned above about neutropenia and lithium ability to reduce the incidence of neutropenia in patient taking chemotherapy without needing to highly costing recombinant granulocyte colony stimulating factors that Egyptian patient can't afford or using the antibiotic as a prophylactic agent that will result in resistance. we want to use lithium to attenuate neutropenia induced chemotherapy. Also because of the anti-cancer activity and neuroprotective properties of lithium that mentioned above we hypothesis that lithium will not conflict with chemotherapy treatment but will help to gain the maximum benefit of chemotherapy and minimize the side effects.

Hypothesis:

Because of the effect of lithium on WBCs and its ability to produce leukocytosis,it is hypothesized that lithium is capable of reversing the chemotherapy induced neutropenia, might be through induction of endogenous colony stimulating factor (CSF) or through alteration of the balance between cytokines that involved in neutrophils mobilization from bone marrow to the blood (CXCl12 and CXCl1).

Aim:

To investigate the efficacy of lithium carbonate in attenuating chemotherapy induced neutropenia, the effect of lithium on granulocyte colony stimulating factor and cytokines involved in neutrophils mobilization from bone marrow to blood in breast cancer patients

Patients and methodology:

This is a prospective randomized study include (50 patients) will be done in collaboration between Clinical Pharmacy Department, Faculty of Pharmacy, Al-Azhar University, Cairo and Clinical Oncology and Nuclear Medicine Department, Faculty of Medicine, Tanta University during June/2020 to June/2021 in breast cancer patients received chemotherapy which induced neutropenia.

ELIGIBILITY:
Inclusion Criteria:

1. All patients presented with breast cancer documented by pathological reports stage I, II and III.

Exclusion Criteria:

1. Patients receiving cardiac medication such as diuretics.
2. Patients on sodium-restricted diet (to avoid lithium toxicity).
3. Stage IV with expected short overall survival.
4. Patients with blood or bone marrow cancer (to prevent interference).
5. Patients with hepatic and renal impairment.
6. Patient with untreated hypothyroidism.
7. Pregnant and breast feeding patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
change in white blood cells count | At baseline (on the 1st day of first cycle) before chemotherapy administration and after each cycle (on the 18th day of every cycle) for six cycles of chemotherapy. (each cycle is 21 days)

SECONDARY OUTCOMES:
G-CSF | At baseline (on the 1st day of first cycle) before chemotherapy administration and after completion of six cycles of chemotherapy (on the 18th day of sixth cycle). (each cycle is 21 days)
CXCL12 | At baseline (on the 1st day of first cycle) before chemotherapy administration and after completion of six cycles of chemotherapy (on the 18th day of sixth cycle). (each cycle is 21 days)
CXCL1 | At baseline (on the 1st day of first cycle) before chemotherapy administration and after completion of six cycles of chemotherapy (on the 18th day of sixth cycle). (each cycle is 21 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University, Cairo, Non-US/Non-Canadian, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bodey GP, Buckley M, Sathe YS, Freireich EJ. Quantitative relationships between circulating leukocytes and infection in patients with acute leukemia. Ann Intern Med. 1966 Feb;64(2):328-40. doi: 10.7326/0003-4819-64-2-328. No abstract available. PMID 5216294
- [Background] el-Mallakh RS. Lithium. Conn Med. 1990 Mar;54(3):115-26. PMID 2182284
- [Background] Slater V, Milanes F, Talcott V, Okafor KC. Influence of age on lithium therapy. South Med J. 1984 Feb;77(2):153-4, 158. doi: 10.1097/00007611-198402000-00003. PMID 6701582
- [Background] Yassa R. Leukocytosis during long-term lithium treatment. N Y State J Med. 1981 Sep;81(10):1479-80. No abstract available. PMID 6792575
- [Background] Ballin A, Lehman D, Sirota P, Litvinjuk U, Meytes D. Increased number of peripheral blood CD34+ cells in lithium-treated patients. Br J Haematol. 1998 Jan;100(1):219-21. doi: 10.1046/j.1365-2141.1998.00537.x. PMID 9450814
- [Background] RADOMSKI JL, FUYAT HN, NELSON AA, SMITH PK. The toxic effects, excretion and distribution of lithium chloride. J Pharmacol Exp Ther. 1950 Dec;100(4:1):429-44. No abstract available. PMID 14804282
- [Background] Petrini M, Vaglini F, Carulli G, Azzara A, Ambrogi F, Bertelli A. Effects of lithium and rubidium on the differentiation of mononuclear cells. Int J Tissue React. 1986;8(5):391-2. PMID 3781770
- [Background] Tisman G, Herbert V, Rosenblatt S. Evidence that lithium induces human granulocyte proliferation: elevated serum vitamin B 12 binding capacity in vivo and granulocyte colony proliferation in vitro. Br J Haematol. 1973 Jun;24(6):767-71. doi: 10.1111/j.1365-2141.1973.tb01704.x. No abstract available. PMID 4716059
- [Background] Harker WG, Rothstein G, Clarkson D, Athens JW, Macfarlane JL. Enhancement of colony-stimulating activity production by lithium. Blood. 1977 Feb;49(2):263-7. PMID 299818
- [Background] Levitt LJ, Quesenberry PJ. The effect of lithium on murine hematopoiesis in a liquid culture system. N Engl J Med. 1980 Mar 27;302(13):713-9. doi: 10.1056/NEJM198003273021303. PMID 6965517
- [Background] Stein RS, Hanson G, Koethe S, Hansen R. Lithium-induced granulocytosis. Ann Intern Med. 1978 Jun;88(6):809-10. doi: 10.7326/0003-4819-88-6-809_2. No abstract available. PMID 666142
- [Background] Kast RE. How lithium treatment generates neutrophilia by enhancing phosphorylation of GSK-3, increasing HIF-1 levels and how this path is important during engraftment. Bone Marrow Transplant. 2008 Jan;41(1):23-6. doi: 10.1038/sj.bmt.1705872. Epub 2007 Oct 1. PMID 17906701
- [Background] Li H, Huang K, Liu X, Liu J, Lu X, Tao K, Wang G, Wang J. Lithium chloride suppresses colorectal cancer cell survival and proliferation through ROS/GSK-3beta/NF-kappaB signaling pathway. Oxid Med Cell Longev. 2014;2014:241864. doi: 10.1155/2014/241864. Epub 2014 Jun 5. PMID 25002914
- [Background] de Araujo WM, Robbs BK, Bastos LG, de Souza WF, Vidal FC, Viola JP, Morgado-Diaz JA. PTEN Overexpression Cooperates With Lithium to Reduce the Malignancy and to Increase Cell Death by Apoptosis via PI3K/Akt Suppression in Colorectal Cancer Cells. J Cell Biochem. 2016 Feb;117(2):458-69. doi: 10.1002/jcb.25294. PMID 26224641
- [Background] Maeng YS, Lee R, Lee B, Choi SI, Kim EK. Lithium inhibits tumor lymphangiogenesis and metastasis through the inhibition of TGFBIp expression in cancer cells. Sci Rep. 2016 Feb 9;6:20739. doi: 10.1038/srep20739. PMID 26857144
- [Background] Zhong Z, Sanchez-Lopez E, Karin M. Autophagy, Inflammation, and Immunity: A Troika Governing Cancer and Its Treatment. Cell. 2016 Jul 14;166(2):288-298. doi: 10.1016/j.cell.2016.05.051. PMID 27419869
- [Background] Sarkar S, Floto RA, Berger Z, Imarisio S, Cordenier A, Pasco M, Cook LJ, Rubinsztein DC. Lithium induces autophagy by inhibiting inositol monophosphatase. J Cell Biol. 2005 Sep 26;170(7):1101-11. doi: 10.1083/jcb.200504035. PMID 16186256
- [Background] Lyman GH, Williams CC, Preston D, Goldman A, Dinwoodie WR, Saba H, Hartmann R, Jensen R, Shukovsky L. Lithium carbonate in patients with small cell lung cancer receiving combination chemotherapy. Am J Med. 1981 Jun;70(6):1222-9. doi: 10.1016/0002-9343(81)90831-7. PMID 6263091